CLINICAL TRIAL: NCT04828772
Title: Real-World Evidence for Anticoagulation Treatment Patterns and Outcomes of Patients Hospitalized With COVID-19 in Japan - A Database Study
Brief Title: A Study of Anticoagulation Treatment Patterns and Outcomes of Participants Hospitalized With Coronavirus Disease 2019 (COVID-19) in Japan
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-801
Record Dates: First submitted 2021-03-25; First posted 2021-04-02 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
Keywords: Anticoagulant; Apixaban; BMS-562247; Coronavirus disease 2019; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cohort 1: COVID-19 participants receiving anticoagulants
- Cohort 2: COVID-19 participants not receiving anticoagulants

SUMMARY:
The purpose of this study is to describe demographic and clinical characteristics of participants who are hospitalized due to coronavirus 2019 (COVID-19), treatment use for COVID-19 and COVID-19 symptoms, and composite outcomes of COVID-19. This study will also compare composite outcomes between COVID-19 participants treated with and without anticoagulant therapy during follow-up period.

ELIGIBILITY:
Inclusion Criteria:

• At least one diagnosis code for COVID-19 (International Classification of Diseases (ICD)-10: U07.1 or B34.2) during hospitalization

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Confirmed COVID-19 patients will be defined as patients who had a diagnosis of COVID-19.Two sub populations will be created based on anticoagulation treatment, and the same outcomes of patient characteristics, treatment patterns and clinical outcomes will be assessed:
  * Sub-population 1: COVID-19 patients receiving anticoagulants
  * Sub-population 2: COVID-19 patients not receiving anticoagulants
Sampling Method: Non-Probability Sample
Enrollment: 9282 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2022-02-07 (Actual)

PRIMARY OUTCOMES:
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Age | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Age group | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Gender | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Index month | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Height | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Weight | At Baseline
Distribution of socio-demographic characteristics of COVID-19 patients who are hospitalized from COVID-19: Body Mass Index (BMI) | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: Treatments | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: Comorbidities | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: Follow-up | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: History of thrombosis | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: Charlson Comorbidity Index (CCI) | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: CCI severity | At Baseline
Distribution of clinical characteristics of COVID-19 patients who are hospitalized from COVID-19: Molecular/diagnosis testing | At Baseline
Distribution of the use of treatments for COVID-19: Anticoagulation | Up to 9 months
Distribution of the use of treatments for COVID-19: Angiotensin-converting enzyme (ACE) inhibitors | Up to 9 months
Distribution of the use of treatments for COVID-19: Angiotensin II receptor blockers (ARBs) | Up to 9 months
Distribution of the use of treatments for COVID-19: ARBs combination | Up to 9 months
Distribution of the use of treatments for COVID-19: Statin | Up to 9 months
Distribution of the use of treatments for COVID-19: HIV protease inhibitor | Up to 9 months
Distribution of the use of treatments for COVID-19: Non-pharmacological treatment | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: Anticoagulation | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: Angiotensin-converting enzyme (ACE) inhibitors | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: Angiotensin II receptor blockers (ARBs) | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: ARBs combinations | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: Statin | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: HIV protease inhibitor | Up to 9 months
Distribution of the use of treatments for COVID-19 symptoms: Non-pharmacological treatment | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: In-hospital death | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: Overall survival | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: Utilization of Extracorporeal membrane oxygenation (ECMO) | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: Utilization of mechanical ventilation (invasive & noninvasive) | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: Utilization of oxygen therapy | Up to 9 months
Distribution of composite outcomes of COVID-19 patients: Intensive care unit/high care unit (ICU/HCU) admission | Up to 9 months

SECONDARY OUTCOMES:
Distribution of composite outcomes of COVID-19 patients treated with anticoagulant therapy during the follow-up period | Up to 9 months
  Severity of COVID-19
Distribution of composite outcomes of COVID-19 patients treated without anticoagulant therapy during the follow-up period | Up to 9 months
  Severity of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- Japan (2):
  - Local Institution, Minato-ku, Tokyo
  - Medical Data Vision, Tokyo

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm